CLINICAL TRIAL: NCT06999798
Title: A Phase 1 Study in Patients With Clinically Node-Positive Breast Cancer to Assess the Safety, Ultrasound Conspicuity, and Migration of an Optimized Ultrasound Twinkling Marker Observed for Sonographic Targeting (UTMOST2 Trial)
Brief Title: An Optimized Ultrasound Twinkling Marker for the Imaging of Lymph Nodes in Patients With Clinically Node-Positive Breast Cancer, The UTMOST2 Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 25-001216; NCI-2025-03536 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-001216 (Other: Mayo Clinic in Rochester); R01EB033008 (NIH)
Record Dates: First submitted 2025-05-16; First posted 2025-05-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Breast Carcinoma
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diagnostic (optimized twinkling marker placement, ultrasound) (Experimental): Patients undergo ultrasound-guided placement of the optimized twinkling marker into the positive lymph node, followed by additional ultrasound imaging and SOC mammography prior to starting NST. Patients also undergo optional ultrasound imaging during NST as clinically indicated. Patients then undergo surgical removal of the optimized twinkling marker during SOC surgical resection of the positive lymph node.
  Interventions: Procedure: Diagnostic Mammography; Procedure: Resection; Procedure: Ultrasound Imaging; Device: Twinkling Marker Placement

INTERVENTIONS:
Procedure: Diagnostic Mammography — Undergo mammography
  Other Names: diagnostic mammogram
Procedure: Resection — Undergo surgical resection of the lymph node as part of standard care.
  Other Names: Surgical Resection
Procedure: Ultrasound Imaging — Undergo ultrasound imaging. Ultrasound images will be evaluated for presence and visibility/conspicuity of the twinkling marker.
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Device: Twinkling Marker Placement — Undergo ultrasound-guided placement of the optimized twinkling marker into the positive lymph node after confirmation of metastatic axillary lymph node involvement.
  Other Names: Twinkle Marker; Mayo Twinkle Marker; Biopsy Twinkle Marker; Biopsy Twinkling Marker; Mayo-designed Twinkling Marker

SUMMARY:
This phase I trial studies the performance, including ultrasound visibility, of an optimized ultrasound twinkling marker in imaging lymph nodes in patients with clinically node-positive breast cancer. In patients with biopsy-proven breast cancer, biopsy markers are used to identify the sites of cancer involvement in both the breasts and lymph nodes. These biopsy markers are critical for guiding surgical management many months after the marker is placed. For breast radiologists and breast surgeons, there is a need for simple, consistent visibility of biopsy markers by ultrasound, particularly several months after marker placement. Ultrasound is the imaging method of choice, particularly for lymph nodes in the armpit (axilla). Ultrasound is non-ionizing and is more comfortable for patients compared to mammography. However, ultrasound visibility of these markers is challenging and inconsistent, with ultrasound failing to detect the marker approximately 25% of the time. The Mayo-designed investigational biopsy marker takes advantage of an ultrasound phenomenon called twinkling artifact. The Mayo-designed optimized ultrasound twinkling marker may work better than standard biopsy clip marker in imaging lymph nodes in patients with clinically node-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older with breast cancer and biopsy-proven malignant involvement of an axillary lymph node
* Surgical management will be determined by the surgeon, who will decide if preoperative Iodine (I)-125 seed localization of the positive node is necessary or if they will retrieve the positive node with intraoperative ultrasound guidance. During surgery, the targeted node, its associated biopsy markers, I-125 seed if placed, and optimized twinkling marker will be resected. The position of the marker in the lymph node or proximity to the node will be noted from the surgical and pathology documentation
* Surgery will be performed by one of the surgeons in the Division of Breast and Melanoma Surgical Oncology (Doctor [Dr.] Judy Boughey, Dr. Amy Degnim, Dr. Tina Hieken, Dr. Jeffrey Johnson, Dr. Mary Mrdutt, Dr. Shon Black)
* Patients must be able to understand the study procedures and comply with them for the entire length of the study
* No contraception is necessary or required

Exclusion Criteria:

* Patients who are pregnant
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Current or past participation within a specified timeframe in another clinical trial, as warranted by the administration of this intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Conspicuity of the optimized Mayo-developed twinkling marker | Baseline up to final pre-operative imaging before surgery; generally 6-9 months
  Assessed by the visibility/conspicuity of the twinkling marker under ultrasound occurring as part of standard of care [neoadjuvant systemic therapy (NST)].
Migration of the optimized Mayo-developed twinkling marker | At time of surgery (baseline)
  Will be determined from surgical and pathology documentation after node resection

SECONDARY OUTCOMES:
Incidence of adverse events (safety of twinkling marker) | Baseline up to final visit before surgery; generally 6-9 months
  Adverse events (AEs) are defined as any untoward or unfavorable medical occurrence in a clinical research study participant, including any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participants' involvement in the research, whether or not considered related to participation in the research. AEs will be assessed as Mild (events require minimal or no treatment and do not interfere with the participant's daily activities); Moderate (events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning); or Severe (Events interrupt a participant's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating).Of note, the term "severe" does not necessarily equate to "serious".

CONTACTS AND LOCATIONS:
Overall Officials: Christine U. Lee, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials